CLINICAL TRIAL: NCT04890093
Title: Phase 1/2 Study of Vincristine and Temozolomide in Combination With PEN-866 for Adolescents and Young Adults With Relapsed or Refractory Solid Tumors
Brief Title: Vincristine and Temozolomide in Combination With PEN-866 for Adolescents and Young Adults With Relapsed or Refractory Solid Tumors
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Pending updated agreements in order to enroll additional participants.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000092; 000092-C
Record Dates: First submitted 2021-05-15; First posted 2021-05-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Sarcoma, Ewing; Rhabdomyosarcoma
Keywords: Sarcoma; Ewing Sarcoma; Rhabdomyosarcoma; Small Molecule
MeSH Terms: conditions — Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma | interventions — Vincristine; Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Dose Escalation (Experimental): Dose escalation of PEN-866 along with fixed doses of vincristine and temozolomide
  Interventions: Drug: PEN-866; Drug: Vincristine; Drug: Temozolomide
- 2/MTD/RP2D (Experimental): PEN-866 at the MTD or RP2D from phase 1 plus vincristine and temozolomide
  Interventions: Drug: PEN-866; Drug: Vincristine; Drug: Temozolomide

INTERVENTIONS:
Drug: PEN-866 — PEN-866 will be given as an IV infusion once every week for the first two consecutive weeks out of every three-week (21 day) cycle.
Drug: Vincristine — Vincristine will be given at a dose of 1.5 mg/m2 by IV on days 1 and 8 of each 21-day cycle
Drug: Temozolomide — temozolomide will be given at a dose of 100 mg/m2, orally on days 1-5, of each 21-day cycle

SUMMARY:
Background:

The drug PEN-866 can remain in tumor cells longer than it does in normal cells. It also may be more effective than other drugs at treating Ewing sarcoma and rhabdomyosarcoma. Researchers want to learn if combining PEN-866 with other drugs can treat certain cancers in adolescents and young adults.

Objective:

To learn if the combination of PEN-866 with vincristine and temozolomide can be used to treat adolescents and young adults with solid tumors that have returned after or did not respond to standard treatments, or for which there are no standard treatments.

Eligibility:

People ages 12-39 years who have solid tumors, Ewing sarcoma, or rhabdomyosarcoma that returned after or did not respond to standard treatments.

Design:

Participants will be screened with a medical history, physical exam, and eye exam. They will have heart function tests. They may have imaging scans of the chest, abdomen, and pelvis. They will give blood and urine samples. They may have a tumor biopsy. Some samples will be used for genetic testing. Some screening tests will be repeated during the study.

Participants will get 3 drugs for up to 18 cycles. Each cycle lasts 21 days. They will get PEN-866 and vincristine by IV infusion (a tube in their vein) on Days 1 and 8 of each cycle. They will take temozolomide by mouth on Days 1-5 of each cycle.

Participants will complete questionnaires about their physical, mental, and social health.

Participants will have a follow-up visit 30 days after treatment ends. They may be contacted by phone or email for the rest of their life.

DETAILED DESCRIPTION:
Background:

Irinotecan is a prodrug of an inhibitor of topoisomerase 1 (active metabolite is SN-38) with known activity in sarcomas, however it has limitations including suboptimal bioavailability and systemic side effects including severe diarrhea and bone marrow suppression.

Preclinical and clinical evidence has demonstrated that prolonged exposure to topoisomerase 1 inhibition produces superior responses in pediatric-type sarcomas, compared to shorter exposures of irinotecan.

PEN-866 is a novel molecule consisting of SN-38 conjugated to a heat shock protein 90 (HSP90) inhibitor that has been shown to have a pharmacokinetic (PK) advantage over irinotecan in preclinical models.

Preclinical and clinical data have shown that PEN-866 acts as a tumor delivery agent for SN-38, allowing SN-38 to remain in tumor cells substantially longer than it remains in normal cells.

In preclinical models of Ewing sarcoma and rhabdomyosarcoma, PEN-866 has superior efficacy and pharmacodynamics compared to irinotecan.

PEN-866 has completed phase 1 testing in adults as a single agent but has yet to be tested in any combinations.

Vincristine/irinotecan/temozolomide (VIT) is a standard relapse regimen for several pediatric sarcomas, with objective responses reported in a subset of participants with Ewing sarcoma and rhabdomyosarcoma.

Objectives:

Phase 1: Determine the maximum tolerated/recommended phase 2 dose (MTD/RP2D) of PEN-866 that can be combined with vincristine and temozolomide in adolescent and young adult (AYA) participants (12-39 years) with relapsed or refractory solid tumors

Phase 2: Determine the objective response rate (CR + PR by RECIST v1.1) of the combination of vincristine, temozolomide and PEN-866 at the RP2D in AYA participants (12-39 years) with relapsed or refractory Ewing sarcoma and rhabdomyosarcoma after a maximum of 18 cycles of the combination

Eligibility:

Phase 1

Age >= 12 and <= 39 years of age

Diagnosis of a relapsed or refractory solid tumor and have archival tissue available.

Adequate performance status and adequate major organ function and have recovered from acute toxicity of all prior therapies.

Phase 2

Age >= 12 and <= 39 years of age

Diagnosis of relapsed or refractory Ewing sarcoma or rhabdomyosarcoma and have archival tissue available

Participants must not have received prior combination therapy with irinotecan and temozolomide

Adequate performance status and adequate major organ function and have recovered from acute toxicity of all prior therapies.

Design:

Open label phase 1/2 study to evaluate the safety and preliminary efficacy of PEN-866 given in combination with vincristine and temozolomide in adolescents and young adults with relapsed or refractory solid tumors

Phase 1 portion will use a standard 3 + 3 design with limited dose escalations to define the MTD or the highest safe dose tested of PEN-866 when given in combination with standard dosing of vincristine (1.5 mg/m2 IV on days 1 and 8) and temozolomide (100 mg/m2 orally on days 1-5) given in 21 day cycles

Phase 2 component will use Simon minimax two-stage phase II trial design and will enroll two expansion cohorts of participants (Ewing sarcoma and rhabdomyosarcoma)

For the Ewing sarcoma cohort, up to a total of 25 evaluable participants will be accrued.

For the rhabdomyosarcoma cohort, up to a total of 17 evaluable participants will be accrued.

A potential additional phase 2 expansion cohort may open for enrollment with an amendment if there are participants with diagnoses other than rhabdomyosarcoma or Ewing sarcoma who have demonstrated possible benefit from this combination by experiencing a response in the phase 1 portion of the trial.

Maximum number of treatment cycles is 18.

A maximum of 12 participants will be required to determine the MTD during phase 1, and a maximum of 42 (25+17) evaluable participants will be accrued for the phase 2 cohorts. To allow for a small number of inevaluable participants and to accommodate screen failures, the accrual ceiling will be set at 64.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Pathology:

  * For phase 1, Participants must have histologically or cytologically confirmed recurrent or refractory solid tumors, excluding CNS tumors and lymphoma.
  * For phase 2, participants must have histologically or cytologically confirmed recurrent or refractory Ewing sarcoma (Cohort 2) or embryonal or alveolar rhabdomyosarcoma (Cohort 3). Participants with Ewing sarcoma (Cohort 2 only) should have evidence of EWS translocation by FISH or RT-PCR.

NOTE: Histologic confirmation of original diagnosis or relapse is required by the Laboratory of Pathology, NCI or participating site s Pathology Department. A formalin fixed tissue block or at least 5 unstained slides (10 micron thick) of archival tumor sample must be available at the time of enrollment. Participants under 18 years old without adequate archival tissue available may opt to undergo pre-treatment biopsy if it can be performed with minimal morbidity. In the event that a participants under 18 cannot safely undergo biopsy and does not have adequate archival tissue available, enrollment will be at the discretion of the Study Chair.

* Measurable disease:

  * For phase 1, participants must have measurable (per RECIST 1.1.) or non-measurable disease on imaging, or presence of recurrent/residual disease identified on aspirate/biopsy or due to presence of elevated tumor biomarkers.
  * For phase 2, participants must have measurable disease, per RECIST 1.1.
* Prior therapy:

  * For phase 1, there are no limits to the number of prior treatment regimens
  * For phase 2, there are no limits to the number of prior treatment regimens. However, participants must not have received any prior therapy with an irinotecan/temozolomide combination containing regimen (participants may have received either drug alone or in combination with different agents at different periods of their course).
  * For all participants: Participants must have recovered from the acute side effects of their prior therapy, such that eligibility criteria are met.

The following prior therapies are permitted, given the indicated time has elapsed:

* Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive. At least 21 days must have elapsed after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea).
* Anti-cancer agents not known to be myelosuppressive (which can include biologic agent, targeted agent, tyrosine kinase inhibitor, or a metronomic non-myelosuppressive regimen): >=7 days must have elapsed after the last dose of agent.
* Antibodies including checkpoint inhibitors: >= 21 days or 3 half-lives (whichever is shorter) must have elapsed from infusion of last dose of antibody.
* Systemic corticosteroids: Participants may be on physiologic steroid replacement for adrenal insufficiency or chronic corticosteroids at a stable dose for at least 7 days. Participants undergoing a steroid wean are eligible as long as no dose re-escalation has occurred in the prior 7 days. If steroids are being used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid, unless the participant is receiving physiologic steroid replacement for adrenal insufficiency.
* Hematopoietic growth factors: >= 14 days after the last dose of a long-acting growth factor (e.g., pegfilgrastim) or 7 days for short-acting growth factor.
* Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days must have elapsed after the completion of dose
* Stem cell infusions (with or without total body irradiation [TBI]):

  * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including DLI or boost infusion: >= 84 days must have elapsed after infusion and no evidence of GVHD.
  * Autologous stem cell infusion including boost infusion: >= 42 days must have elapsed.
  * Cellular Therapy: >= 42 days must have elapsed after the completion of any type of cellular therapy (e.g., modified T cells, NK cells, dendritic cells, etc.).
* XRT/External Beam Irradiation including Protons: >= 84 days after TBI, craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow radiation. >= 14 days after local XRT however there is no time restriction for palliative radiation with minimal bone marrow involvement and the participant has measurable/evaluable disease outside the radiation port or the site of radiation has documented progression.
* Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days must have elapsed after systemically administered radiopharmaceutical therapy.

  * Age >= 12 years and <= 39 years

NOTE: Because no dosing or adverse event data are currently available on the use of PEN-866 in participants <18 years of age, children <12 years of age are excluded from this study but will be eligible for future pediatric trials. Since the study population of interest is relapsed or refractory sarcomas which is typically seen in adolescents and young adults, and per FDA recommendations for enrolling adolescents in disease/target-appropriate adult oncology clinical trials of investigational agents, eligibility will include participants aged 12-17 years old.

* ECOG performance status <=2, (Karnofsky >=50% for participants > 16 years of age and Lansky >= 50% for participants <= 16 years of age. NOTE: Neurologic deficits in participants with CNS metastases must have been stable for at least 7 days prior to study enrollment. Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of performance.
* Willingness to have a central venous access line placed if the participant does not already have one in place.
* Participants must have adequate organ and marrow function as defined below:

Hematologic Function:

* Peripheral absolute neutrophil count (ANC) >= 1000/mm3
* Platelet count >=75,000/mm^3
* Hemoglobin >= 8 g/dL

  * Participants without known metastatic bone marrow disease must meet the blood counts as listed above, without requiring transfusions (defined as not receiving platelet or red blood cell transfusions for at least 7 days prior to initiation of study therapy) or growth factor support
  * For participants with known metastatic bone marrow disease:

    * Provided they meet the blood counts as listed above, without requiring transfusions (defined as not receiving platelet or red blood cell transfusions for at least 7 days prior to initiation of study therapy) or growth factor support these participants will be eligible for the phase 1 component of the study.
    * For the phase 2 component, participants should meet the blood counts as listed above, but may receive transfusions of red blood cells or platelets provided they are not known to be refractory to red cell or platelet transfusions. These participants will be excluded from the phase 1 component.
  * For participants undergoing biopsy only, adequate coagulation defined as INR <= 1.5

Renal Function:

* Creatinine clearance or radioisotope GFR >= 60 mL/min/1.73 m^2 or
* A serum creatinine based on age/gender as follows:

Age 12 to <13 years maximum serum creatine male 1.2 female 1.2

Age 13 to <16 years maximum serum creatine male 1.5 female 1.4

Age >= 16 years maximum serum creatine male 1.7 female 1.4

The Cockcroft-Gault equation should be used for calculation of creatinine clearance.

Liver Function:

* Bilirubin (sum of conjugated + unconjugated) <= 1.5 upper limit of normal (ULN) for age
* SGPT (ALT) <= 135 U/L.
* SGOT (AST) <= 150 U/L.

Participants with Gilbert s syndrome are excluded from the requirement of a normal bilirubin unless they are found to have the UGT1A1 28/28 genotype. Gilbert s syndrome is found in 3-10% of the general population, and is characterized by mild, chronic unconjugated hyperbilirubinemia in the absence of liver disease or overt hemolysis. NOTE: Adult values will be used for calculating hepatic toxicity and determining eligibility.

Cardiac Function:

* Shortening fraction of >=27% or ejection fraction of >= 50% by echocardiogram.
* QTc interval < 470 msec

  * Participants with toxicities from prior therapies must have resolution of these toxicities to <= Grade 1, with the exception of peripheral neuropathy and alopecia which must resolve to <=Grade 2.
  * Participants with treated brain metastases (CNS as primary tumor not eligible) are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression. Participants must be asymptomatic from their brain metastasis and not require corticosteroids for 4 weeks prior to start of therapy (C1D1). Participants with remote history of spinal cord compression are eligible.
  * Participants with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy. Participants must be asymptomatic or have disease controlled with surgery and radiation and should not require steroids within 4 weeks prior to start of therapy (C1D1).
  * Participants with human immunodeficiency virus (HIV)-infected participants on effective anti- retroviral therapy with no detectable viral load on any tests within the last 6 months are eligible for this trial
  * For participants with chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy within the last 6 months.
  * Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load within the last 6 months.
  * Participants ages 18 years old and older must be willing to undergo tumor biopsy before treatment and have available archival tissue (specifically, a formalin fixed tissue block or at least 5 unstained slides [10 micron thick]) at the time of enrollment. If biopsy is contraindicated or unable to be performed and/or there is no archival tissue available, enrollment must be approved by the Study Chair.
  * Participants ages 12-17 years old without available archival tissue (specifically, a formalin fixed tissue block or at least 5 unstained slides [10 micron thick]) at the time of enrollment may opt to undergo pre-treatment biopsy if it is clinically indicated or if it can be performed with minimal morbidity using local anesthesia. In the event that a participant 12-17 cannot undergo biopsy as described above and does not have adequate archival tissue available, enrollment will be at the discretion of the Study Chair.
  * Individuals of childbearing potential: negative serum Beta human chorionic gonadotropin ((Beta)hCG) pregnancy test during screening. A negative pregnancy test is also required within 8 days before first treatment; screening results may be used for treatment if they fall within the required window.
  * Participants of reproductive potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time of consent, for the duration of therapy, and for 6 months after the last dose of study therapy.
  * Nursing participants must be willing to discontinue nursing from study treatment initiation through 6 months after completion of chemotherapy
  * Ability of participant (or parent or legal guardian in case of pediatric participant) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Participants who are receiving any other investigational agents or other anticancer agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PEN-866 (which includes ganetespib or other HSP90 inhibitors, irinotecan, SN-38, or other agents containing irinotecan, SN-38 or its derivatives) or other agents used in study (vincristine and temozolomide).
* Participants who have previously discontinued vincristine, temozolomide, or irinotecan due to severe toxicity.
* Participants with a history of grade 4 vincristine-related peripheral neuropathy or constipation.
* Participants who require medication with any of the inhibitors of UGT1A1, substrates of CYP1A2 or substrates of the P-gp, BCRP, OATP1B1, OATP1B3, or OCT1 transporters. Participants discontinuing these drugs must undergo a washout of 2-weeks or 5 half-lives, whichever is shorter, prior to C1D1.
* Uncontrolled intercurrent illness as listed below:

  * Unstable angina within 6 months prior to start of treatment
  * Myocardial infarction within 6 months prior to start of treatment
  * New York Heart Association Class III - IV heart failure
  * Clinically important abnormalities in rhythm, conduction, or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block)
  * Congenital long QT syndrome
  * Uncontrolled hypertension despite use of antihypertensives for management of hypertension
  * Stroke or transient ischemic attack within 6 months prior to start of treatment
  * As judged by the investigator, evidence of severe or uncontrolled systemic disease, active bleeding diatheses, renal or liver transplant, or Grade >2 active infection
  * Any medical, psychological, or social condition that would interfere with the participant s participation in the study.
  * Any other uncontrolled intercurrent systemic illness that would limit compliance with study requirements
* Pregnancy
* Major surgery within 28 days prior to start of therapy (C1D1)
* UGT1A1 Status

Participants identified with a UGT1A1 28/28 genotype will be excluded from the phase 1 component of the study. In phase 2, they may receive PEN-866 with altered dosing- see Section. Participants who are known to not be homozygous for UGT1A128/28 genotype (i.e., 1/1 or 1/28) may receive the enrolling cohort dose level of PEN-866 on C1D1 during phase 1 and the RP2D of PEN-866 during phase 2.

Ages: 12 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Objective response rate | baseline to 18 cycles
  complete response + partial response
Phase 1: Maximum tolerated/recommended phase 2 dose | baseline to 18 cycles
  toxicity type/grade and the fraction of patients with a DLT at each dose level

SECONDARY OUTCOMES:
Phase 1: Plasma and tumor pharmacokinetics | pre/post infusion on Cycle 1 Day 1, 24 hr post infusion, Cycle 1 Day 4, Cycle 1 Day 8. Cycle 3 Day 1 and Cycle 3 day 8
  Descriptive report of plasma and tumor pharmacokinetics (PK) of PEN-866 in combination with vincristine and temozolomide
Phase 1: Toxicity | baseline to 18 cycles
  Incidence of specific toxicities
Phase 2: Progression free survival | from start of treatment to time of progression or death
  Median amount of time subject survives without disease progression after treatment
Phase 2: Duration of response | baseline to 18 cycles
  Duration from the date a response is identified until the date of progression or date the response is noted to have ended
Phase 2: Phospho-gamma-H2AX immunofluorescence | Cycle 1 day 1 and Cycle 1 day 4
  Levels of phospho-gamma-H2AX immunofluorescence in matched pre- and on-treatment tumor and normal tissue (hair follicle)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Heske, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000092-C.html